CLINICAL TRIAL: NCT07136012
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study Assessing Olpasiran Use to Prevent First Major Cardiovascular Events in Participants With Elevated Lipoprotein(a)
Brief Title: OCEAN(a)-PreEvent - Olpasiran Trials of Cardiovascular Events And LipoproteiN(a) Reduction to Prevent First Major Cardiovascular Events
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230222
Expanded Access: NCT07079267 (Available)
Record Dates: First submitted 2025-08-18; First posted 2025-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Disease
Keywords: Olpasiran; AMG 890; Coronary heart disease; CHD; Myocardial infarction; Coronary revascularization
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction | interventions — olpasiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olpasiran (Experimental): Participants will receive subcutaneous (SC) olpasiran.
  Interventions: Drug: Olpasiran
- Placebo (Placebo Comparator): Participants will receive SC placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olpasiran — Olpasiran will be administered via SC injection.
  Other Names: AMG 890
  Arms: Olpasiran
Drug: Placebo — Placebo will be administered via SC injection.
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the effect of olpasiran, compared to placebo, on the risk for coronary heart disease death (CHD death), myocardial infarction, or urgent coronary revascularization in participants at risk for a first major cardiovascular event with elevated lipoprotein(a) (Lp[a]).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Lp(a)≥ 200 nmol/L during screening
* Multiple atherosclerotic cardiovascular disease risk factors, and/or evidence of atherosclerosis

Exclusion Criteria:

* Prior acute atherothrombotic event (myocardial infarction, stroke, transient ischemic attack, acute limb ischemia)
* Prior or planned arterial revascularization
* History of major bleeding disorder

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2031-10-20 (Estimated); Study Completion 2031-10-20 (Estimated)

PRIMARY OUTCOMES:
Time to CHD Death, Myocardial Infarction, or Urgent Coronary Revascularization, Whichever Occurs First | Up to approximately 6.2 years

SECONDARY OUTCOMES:
Time to Cardiovascular Death, Myocardial Infarction, or Ischemic Stroke, Whichever Occurs First | Up to approximately 6.2 years
Time to Cardiovascular Death, Myocardial Infarction, Urgent Coronary Revascularization, or Ischemic Stroke, Whichever Occurs First | Up to approximately 6.2 years
Percent Change From Baseline to Week 48 Lp(a) Levels | Baseline and Week 48
Time to Myocardial Infarction | Up to approximately 6.2 years
Time to CHD Death or Myocardial Infarction, Whichever Occurs First | Up to approximately 6.2 years
Time to Urgent Coronary Revascularization | Up to approximately 6.2 years
Time to Coronary Revascularization | Up to approximately 6.2 years
Time to CHD Death | Up to approximately 6.2 years
Time to Cardiovascular Death | Up to approximately 6.2 years
Time to Death by any Cause | Up to approximately 6.2 years
Time to Ischemic Stroke | Up to approximately 6.2 years
Serum Concentration of Olpasiran | Up to Week 48
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to approximately 6.2 years
  Including serious adverse events and adverse events leading to discontinuation of investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (215):
- United States (177):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - University of Alabama Birmingham Saint Vincents Birmingham, Birmingham, Alabama
  - Alliance For Multispecialty Research - Daphne, Daphne, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - CB Flock Research Corporation, Mobile, Alabama
  - Phoenix Clinical, Phoenix, Arizona
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - Hero Clinical Research, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - National Heart Institute, Beverly Hills, California
  - 310 Clinical Research, Inglewood, California
  - University of California San Diego, La Jolla, California
  - InvivoCure, Los Angeles, California
  - Valley Clinical Trials, Northridge, California
  - Clinical Trials Research - Sacramento, Roseville, California
  - Alliance Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Manshadi Heart Institute, Stockton, California
  - Blue Coast Cardiology, Vista, California
  - Diablo Clinical Research, Walnut Creek, California
  - Focus Clinical Research, West Hills, California
  - UCHealth Memorial Central, Colorado Springs, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Proactive Clinical Research, Fort Lauderdale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Lake City, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Inpatient Research Clinic, LLC, Miami Lakes, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Eminat, LLC, Miramar, Florida
  - Suncoast Clinical Research Inc, New Port Richey, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Baptist Health Care, Pensacola, Florida
  - Denali Health Plant City, Plant City, Florida
  - FWD Clinical Research, Tamarac, Florida
  - Guardian Research Organization LLC, Winter Park, Florida
  - Emory University Hospital, Atlanta, Georgia
  - East Coast Institute for Research, Canton, Georgia
  - Northeast Georgia Medical Center Wisteria Building, Cumming, Georgia
  - Nsc Research, Johns Creek, Georgia
  - Georgia Clinical Research, Lawrenceville, Georgia
  - St Lukes Idaho Cardiology Associates, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Christie Clinic, Champaign, Illinois
  - Alliance for Multispecialty Research, LLC - Park Ridge, Park Ridge, Illinois
  - MediSphere Medical Research Center LLC, Evansville, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Heart Center, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - Hutchinson Clinic PA, Hutchinson, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Heart Clinic of Hammond, Covington, Louisiana
  - Ima Clinical Research, Monroe, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Monroe Research LLC, West Monroe, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants LLC, Beltsville, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Flourish Research, Bowie, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Centennial Medical Group, Columbia, Maryland
  - Medstar Franklin Square Medical Center, Hyattsville, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - MyMichigan Medical Center Midland - Clinical Research Department, Midland, Michigan
  - Advanced Cardiology Associates, Rochester Hills, Michigan
  - Revival Research Institute, Southfield, Michigan
  - Health East Cancer Care, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Sisters of Saint Mary Health Heart and Vascular Care, Bridgeton, Missouri
  - Washington University, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - American Institute of Medical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Renown Institute for Heart and Vascular Health, Reno, Nevada
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Clinical Reseach Philadelphia Pennington, Hamilton, New Jersey
  - Med Clinical Research Partners - Irvington, Irvington, New Jersey
  - New Jersey Medcare / New Jersey Heart, Linden, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - Circuit Clinical / Optum Medical Care of New Jersey, Secaucus, New Jersey
  - The Heart House - Washington Township, Sewell, New Jersey
  - CardioMetabolic Collaborative Clinic, Somerset, New Jersey
  - Ima Clinical Research - Warren, Warren Township, New Jersey
  - Albany Medical College, Albany, New York
  - Basil Clinical, Inwood, New York
  - Rasai Research, Jackson Heights, New York
  - Crystal Run Healthcare, Monroe, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ima Clinical Research Manhattan, New York, New York
  - Niagara Falls Memorial Medical Center, Niagara Falls, New York
  - Circuit Clinical Orchard Park Family Practice, Orchard Park, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Accellacare Research of Wilmington, Wilmington, North Carolina
  - Aultman Cardiology Clinical Trials, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Nexgen Research, Lima, Ohio
  - K and R Research, Marion, Ohio
  - Alliance for Multispecialty Research, Norman, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pottstown Medical Specialists Inc, Pottstown, Pennsylvania
  - Pharmacorp Clinical Trials Inc, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Carolina Cardiology - Greenville, Gantt, South Carolina
  - Walker Family Care, Little River, South Carolina
  - Accellacare Charleston, Mt. Pleasant, South Carolina
  - Tribe Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Erlanger Health, Inc., Chattanooga, Tennessee
  - Apex Research Foundation, LLC, Jackson, Tennessee
  - Alliance for Multispecialty Research Knoxville, Knoxville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Ima Clinical Research, Austin, Texas
  - Pioneer Medical Associates, Carrollton, Texas
  - Baylor Scott and White Heart and Vascular Hospital-Dallas, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Cedar Health Research, LLC, Dallas, Texas
  - Cedar Health Research, LLC, Euless, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Cardiovascular Specialists of Willowbrook, Houston, Texas
  - Vital Heart and Vein, Humble, Texas
  - Tcr Institute Llc, Kingwood, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Orion Medical, Pasadena, Texas
  - Valley Institute of Research Plano, Plano, Texas
  - Ima Clinical Research San Antonio, San Antonio, Texas
  - St Davids Heart & Vascular PLLC dba Austin Heart, San Marcos, Texas
  - Revival Research Institute, Sherman, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Alpine Research Organization, Layton, Utah
  - Inova Cardiology - Fairfax, Fairfax, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Newport News, Virginia
  - Alliance for Multispecialty Research Norfolk, Norfolk, Virginia
  - Centricity Research, Suffolk, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Western Washington Medical Group, Everett, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Australia (20):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Novatrials, Charlestown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Aim Research, Merewether, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Advara HeartCare Wesley, Auchenflower, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - University of The Sunshine Coast Clinical Trials, Sippy Downs, Sippy Downs, Queensland
  - Dr Heart Pty Ltd, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Fusion Clinical Research, Norwood, South Australia
  - Victorian Heart Hospital, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Momentum Clinical Research - Sunshine, Melbourne, Victoria
  - Clinitrials - Mandurah, Greenfields, Western Australia
  - Advara HeartCare Joondalup, Joondalup, Western Australia
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia
  - Clinitrials - Mount Medical Centre, Perth, Western Australia
- Canada (18):
  - Centricity Research Calgary, Calgary, Alberta
  - Edmonton Cardiology Consultants, Edmonton, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - SMH Cardiology Clinical Trials Incorporated, Surrey, British Columbia
  - ARC Biosystems Incorporated, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Discovery Clinical Services Ltd, Victoria, British Columbia
  - Centricity Research Brampton, Brampton, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - Elevate Clinical Research KMH Missisauga, Mississauga, Ontario
  - Partners in Advanced Cardiac Evaluation, Newmarket, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Institut de recherches cliniques de Montreal, Montreal, Quebec
  - Research Institute of McGill University Health Center - Glen Site, Montreal, Quebec
  - CIUSSS de l Estrie CHUS Hopital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com